CLINICAL TRIAL: NCT01195051
Title: Medication Reconciliation Technology to Improve Quality of Transitional Care
Acronym: MedMatch
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Regenstrief Institute, Inc. (Other); Wishard Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0910-19; R18HS018183 (AHRQ)
Record Dates: First submitted 2010-07-12; First posted 2010-09-03 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Medication Reconciliation
Keywords: Medication Reconciliation; Inpatient; Electronic Medical Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electronic medication reconciliation (Experimental): Providers have access to a new, computer-based application to facilitate documentation and prescribing of outpatient medications in the inpatient setting.
  Interventions: Other: Electronic medication reconciliation
- Control (No Intervention)

INTERVENTIONS:
Other: Electronic medication reconciliation — A new, computer-based application will be used to document and prescribe outpatient medications in the inpatient setting.
  Other Names: MedMatch
  Arms: Electronic medication reconciliation

SUMMARY:
This study addresses the problem of inadequate medication reconciliation as patients cross boundaries between inpatient and outpatient care (ambulatory care). The purpose of this study is to determine whether a new, computer-based application, integrated with electronic prescribing, improves erroneous discrepancies between pre-hospital medications and medications upon patients' return to ambulatory care.

DETAILED DESCRIPTION:
This project will test a systems-based intervention of the electronic medical records system. The specific aims of this study are to integrate a new electronic medication reconciliation (MR) system with an electronic prescribing system, conduct a randomized controlled trial of MR, and determine whether electronic facilitation of MR alters MR and the incidence of medication errors in ambulatory care. On a patient's hospital admission, a new Web-based MR module will receive an automatically compiled outpatient medication list. Following discussion with the patient, medical personnel will update the list, which will then be delivered to the computer-based provider order entry system and become actionable for prescribing. Main outcomes include adverse drug events and erroneous discrepancies between the pre-admission medication list and the medication list upon the patient's return to ambulatory care. We hypothesize that electronic facilitation of inpatient MR will improve completion of MR and will decrease the incidence of drug-related medical errors.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Medicine Service during a 12-month period
* Physicians who provide inpatient or ambulatory care for participating patients.
* Pharmacists who provide care for participating patients.

Exclusion Criteria:

* Patients admitted but not seen in a primary-care clinic within the preceding 12 months
* If an enrolled subject is determined to be a prisoner or pregnant woman, then the study will discontinue the subject for research purposes or will submit an amendment at that time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4818 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Reconciliation of outpatient medications | Hospital admission, transfer, and discharge; 1 year
  Number and fraction of outpatient medications prescribed or addressed as to why prescribing did not occur. Number and fraction of cases with MR by a pharmacist. Number and fraction of cases undergoing any MR. Number and fraction of cases where any outpatient medications were not prescribed or addressed as to why prescribing did not occur.

SECONDARY OUTCOMES:
Measurement of potential for harm and potential severity of harm | Hospital discharge; 1 year
  For each medication discrepancy, the study team will reach consensus about potential for harm and potential severity of harm. The study team will adopt the following framework: little or no confidence (e.g., omission of multivitamin); slight to modest confidence (e.g., docusate 200 mg every morning, instead of 100 mg twice daily); less than 50% chance but close call (e.g., omission of as-needed enema at discharge); more than 50% chance but close call (e.g., omission of fluticasone twice daily at discharge); or strong confidence (e.g., omission of as-needed haloperidol).
Measurement and analysis of providers' perspectives | Start and end of trial; 1 year
  We will conduct a before-and-after survey of providers. Providers will be surveyed about satisfaction with care, managing medications, and usefulness of local information systems in managing medications.
Measurement and analysis of patients' perspectives | Hospital discharge; 1 year
  The inpatient geriatrics consultation service has begun calling patients who received geriatrics consultation and were subsequently discharged to home. The calls are made by telephone within 72 hours of discharge. Patients are asked eight to ten questions, addressing satisfaction with care, receipt of information about medications, and adherence to medications.
Reportable financial and organizational dimensions | Start of trial; time 0 and 1 year
  We will track and report hours required for several parts of the development and implementation, as follows: hours required for new technical development; and hours providers spend in learning about system and how to use it.
Utilization of intervention | Hospital admission, transfer, and discharge; 1 year
  Fraction of intervention admissions for which Web-based medication list was reviewed or modified. Mean duration of use of Web-based application. Fraction of intervention admissions, transfers, and discharges for which new medication list was used to order medications. Fraction of medications on medication list that were ordered on admission, transfer, and discharge. Timing of when medication reconciliation occurred.
Measurement and analysis of drug-related medical errors | Hospital discharge; 1 year
  At discharge, we will assess for unintentional medication discrepancies at discharge. At ambulatory followup, we will assess whether the medications should have been prescribed at discharge. When a patient is discharged from the hospital and resumes ambulatory care, the patient is expected to adhere to the discharge prescriptions. Each discharge will be reviewed by members of the study team, to determine, for each medication listed on the pre-admission medication list but not prescribed at discharge, whether the discrepancy was intentional or unintentional.
Measurement of adverse drug events and near misses | Hospital discharge; 1 year
  We will count deaths and will identify and assess adverse drug events (ADEs). The following kinds of triggers will be used to identify encounters that might reflect ADEs: diagnostic codes for diagnoses associated with ADEs, potential ADEs, or medication errors; use of specific drugs suggesting that an ADE may have occurred; potentially dangerous drug combinations; combinations of drugs and symptoms (e.g., angiotensin converting enzyme inhibitor and cough); combinations of diagnoses and drugs; and combinations of drugs and miscellaneous.
Medication discrepancies between pre-admission and ambulatory followup | Ambulatory followup; 18 months
  Mean number of erroneous discrepancies between pre-admission and ambulatory followup

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weiner, MD, MPH, Principal Investigator — Indiana University School of Medicine, Department of Medicine
Locations (1):
- Wishard Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Cadwallader J, Spry K, Morea J, Russ AL, Duke J, Weiner M. Design of a medication reconciliation application: facilitating clinician-focused decision making with data from multiple sources. Appl Clin Inform. 2013 Mar 13;4(1):110-25. doi: 10.4338/ACI-2012-12-RA-0057. Print 2013. PMID 23650492